CLINICAL TRIAL: NCT02102100
Title: Menthol's Effects on Nicotine Reinforcement in Smokers
Brief Title: The Effects of Menthol as Delivered by an Electronic Cigarette on the Desirability of Nicotine in Tobacco Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1309012678; 1P50DA036151-01 (NIH)
Record Dates: First submitted 2013-10-07; First posted 2014-04-02 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Nicotine Dependence
Keywords: menthol, electronic cigarette, nicotine, smoking, tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Smoking | interventions — Nicotine; Menthol

STUDY DESIGN:
Intervention Model Description: Subjects in each of the 2 arms received a random sequence of 3 different inhaled menthol conditions across 3 test sessions (a single menthol condition for each test session). In each test session, a random order of one saline, and 2 nicotine (0.25 mg and 0.5 mg /70 kg) infusions were given one hour apart, concurrent with the randomized menthol inhalation condition for that test session. The randomized sequence of nicotine infusions was the same for each test session.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Menthol-Preferring Smokers (Experimental): Each subject in this arm received a random sequence of 3 different inhaled menthol conditions across 3 test sessions (a single menthol condition for each test session). In each test session, a random order of one saline, and 2 nicotine (0.25 mg and 0.5 mg /70 kg) infusions were given one hour apart, concurrent with the randomized menthol inhalation condition for that test session.
  Interventions: Drug: nicotine; Drug: menthol
- Non-Menthol Preferring Smokers (Experimental): Each subject in this arm received a random sequence of 3 different inhaled menthol conditions across 3 test sessions (a single menthol condition for each test session). In each test session, a random order of one saline, and 2 nicotine (0.25 mg and 0.5 mg /70 kg) infusions were given one hour apart, concurrent with the randomized menthol inhalation condition for that test session.
  Interventions: Drug: nicotine; Drug: menthol

INTERVENTIONS:
Drug: nicotine — In each of 3 test sessions, subjects in each arm will receive a randomized sequence of three intravenous infusions (30 sec each), one hour apart. The infusions will consist of saline, nicotine (.25 mg / 70kg) and nicotine (0.5 mg / 70 kg). The randomized sequence will remain the same between test sessions for a given subject.
Drug: menthol — In each of 3 test sessions, subjects will take 6 inhalations from the study e-cigarette, one inhalation every 15 seconds, of the randomized menthol condition for that test session ust prior to each intravenous infusion. The menthol conditions are: 3.2% menthol, 0.5% menthol and tobacco-flavor only (0.0% menthol)
  Other Names: racemic menthol

SUMMARY:
This study will help determine if menthol administered by inhalation via electronic cigarettes (e-cigarette) changes the reinforcing effects of pure nicotine administered intravenously in cigarette smokers who smoke mentholated or non-mentholated cigarettes.

DETAILED DESCRIPTION:
Male and female smokers will be recruited from the New Haven area through newspaper advertisements, radio advertisements, and fliers. Interested subjects will have the study described over the telephone, and they will be asked to answer a brief tobacco use history and medical screening questionnaire. If subjects pass the telephone screening, they will be invited to come to the West Haven VA clinic for a screening evaluation. This screening evaluation will be for the menthol / nicotine reinforcement study as described in detail in this project description. The dose-finding study was conducted at the John B. Pierce Laboratory. The dose finding study concluded with the establishment of the high and low dose of menthol that will be used in this protocol "Menthol's Effects on Nicotine Reinforcement in Smokers." The screening of these subjects used the same inclusion and exclusion criteria as described below.

Inclusion criteria: Female and male smokers, aged 18 to 30 years; history of smoking for the past 12 months, at least one cigarette per day; smoking status is verified with urinary cotinine levels above 10 ng/ml; not seeking treatment for nicotine dependence at the time of study entry; in good health as verified by medical history, screening examination, and screening laboratory tests; for women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion criteria: History of major medical illnesses that the physician investigator deems as contraindicated for the patient to be in the study; regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics); psychiatric diagnosis and / or treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia or panic disorder in the past month and abuse of alcohol or any other recreational or prescription drugs in the past 30 days. Any allergy to propylene glycol or menthol.

This outpatient, double-blind, placebo-controlled study consisted of an adaptation session followed by three test sessions. All participants were randomized to a test session order and received control menthol (0.0% + tobacco flavor), low menthol (0.5% + tobacco flavor), and high menthol (3.2% + tobacco flavor) by standardized inhalation from an e-cigarette just prior to each nicotine infusion (a single menthol condition for each test session). Within each test session, all 3 IV nicotine conditions were tested, one hour apart, by delivering saline, nicotine at 0.25 mg nicotine/70 kg and nicotine at 0.5 mg nicotine/70 kg, in a random order, just after last inhalation. For each participant, the randomized nicotine infusion sequence was fixed across the three test sessions, each performed at least 24 hours apart.

ELIGIBILITY:
Inclusion Criteria:

* Female and male smokers, aged 18 to 30 years;
* History of smoking for the past 12 months, at least one cigarette per day; smoking status is verified with urinary cotinine levels above 10 ng/ml;
* Not seeking treatment for nicotine dependence at the time of study entry;
* In good health as verified by medical history, screening examination, and screening laboratory tests;
* For women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

* History of major medical illnesses that the physician investigator deems as contraindicated for the patient to be in the study
* Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics);
* A psychiatric diagnosis and / or treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia or panic disorder in the past month
* Abuse of alcohol or any other recreational or prescription drugs in the past 30 days.
* Any allergy to propylene glycol or menthol.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, MD, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut VA Healthcare System, West Haven, Connecticut
  - VA Connecticut Health Care System, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female smokers between the ages of 18 and 30 yrs, with a history of smoking for the past 12 months, at least one cigarette per day.
Groups:
- Menthol-Preferring Smokers; Non-Methol Preferring Smokers: Each subject in this arm received a random sequence of 3 different inhaled menthol conditions across 3 test sessions (a single menthol condition for each test session). In each test session, a random order of one saline, and 2 nicotine (0.25mg and 0.5mg/70kg) infusions were given one hour apart, concurrent with the randomized menthol inhalation condition for that test session.
Period: Overall Study
Arm/Group | Menthol-Preferring Smokers | Non-Methol Preferring Smokers
Started | 32 | 25
Completed | 23 | 18
Not Completed | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Menthol-Preferring Smokers: Menthol smokers randomized to a test session order and received control menthol (0.0% + tobacco flavor), low menthol (0.5% + tobacco flavor), and high menthol (3.2% + tobacco flavor) by standardized inhalation from an e-cigarette just prior to each nicotine infusion (a single menthol condition for each test session). Within each test session, all three IV nicotine conditions were tested, 1 hour apart, by delivering saline, nicotine at 0.25 mg nicotine/70 kg and nicotine at 0.5 mg nicotine/70 kg, in a random order, just after last inhalation. For each participant, the randomized nicotine infusion sequence was fixed across the three test sessions, each performed at least 24 hours apart.
- Non-Menthol-Preferring Smokers: Non-menthol smokers randomized to a test session order and received control menthol (0.0% + tobacco flavor), low menthol (0.5% + tobacco flavor), and high menthol (3.2% + tobacco flavor) by standardized inhalation from an e-cigarette just prior to each nicotine infusion (a single menthol condition for each test session). Within each test session, all three IV nicotine conditions were tested, 1 hour apart, by delivering saline, nicotine at 0.25 mg nicotine/70 kg and nicotine at 0.5 mg nicotine/70 kg, in a random order, just after last inhalation. For each participant, the randomized nicotine infusion sequence was fixed across the three test sessions, each performed at least 24 hours apart.
- Total: Total of all reporting groups
Arm/Group | Menthol-Preferring Smokers | Non-Menthol-Preferring Smokers | Total
Number analyzed (Participants) | 32 | 25 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 25 | 57
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.2 (3.6) | 24.0 (3.6) | 24.1 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 1 | 13
  Male | 20 | 24 | 44
Region of Enrollment [Number; unit: participants]
  United States | 32 | 25 | 57
Nicotine Metabolite Ratio [Mean (Standard Deviation); unit: ratio] — Ratio of plasma 3'-hydroxycotinine / cotinine at baseline
  ratio | 0.29 (0.19) | 0.55 (0.35) | 0.40 (.30)

OUTCOME MEASURES:

1. Primary Outcome: Drug Effects Questionnaire (DEQ)- 'Good Drug Effects'
Description: The Drug Effects Questionnaire (DEQ) is used in studies of acute subjective response (SR) to a variety of substances. The DEQ consists of 11 questions: cooling effect, dislike the sensation, any sensations, feel a drug effect, high, feel stimulated, feel a head rush, like drug effect, dislike any effects, craving a cigarette, and like more of the drug. To calculate the DEQ- 'Good Drug Effects', peak values from post-infusion time points were calculated for the change in the intensity of positive subjective effects as measured with 2 DEQ questions - DEQ question #6 'like drug effect' and DEQ question #11 'would like more of the drug'. Each question was measured on a scale with a minimum score of 0 and a maximum score of 100.The peak values for "like" and " I want more" were averaged to obtain a summary score to represent the feel 'Good Drug Effects' composite factor. DEQ measures were skewed and square root transformations were used. Higher scores indicate more positive effects.
Time Frame: up to 55 minutes post-infusion
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Menthol-Preferring Smokers; Non-Menthol Preferring Smokers: Each subject in this arm received a random sequence of 3 different inhaled menthol conditions across 3 test sessions (a single menthol condition for each test session). In each test session, a random order of one saline, and 2 nicotine (0.25 mg and 0.5 mg /70 kg) infusions were given one hour apart, concurrent with the randomized menthol inhalation condition for that test session.
  nicotine: In each of 3 test sessions, subjects in each arm will receive a randomized sequence of three intravenous infusions (30 sec each), one hour apart. The infusions will consist of saline, nicotine (.25 mg / 70kg) and nicotine (0.5 mg / 70 kg). The randomized sequence will remain the same between test sessions for a given subject.
  menthol: In each of 3 test sessions, subjects will take 6 inhalations from the study e-cigarette, one inhalation every 15 seconds, of the randomized menthol condition for that test session ust prior to each intravenous infusion. The menthol conditions are: 3.2% menthol, 0
Arm/Group | Menthol-Preferring Smokers | Non-Menthol Preferring Smokers
Number analyzed (Participants) | 32 | 25
scores on a scale
  Across Conditions (main effect) | 5.1979 (0.3803) | 6.8384 (0.4292)
  High Menthol w High Nicotine | 5.6235 (0.4731) | 7.6285 (0.5287)
  High Menthol w Low Nicotine | 5.226 (0.4766) | 7.4351 (0.5302)
  High Menthol w Saline | 5.0699 (0.4768) | 7.6285 (0.5287)
  Low Menthol w High Nicotine | 5.8971 (0.4736) | 7.5808 (0.5346)
  Low Menthol w Low Nicotine | 5.5481 (0.4809) | 6.7656 (0.5363)
  Low Menthol w Saline | 4.4655 (0.4741) | 6.3960 (0.5307)
Statistical Analysis 1: Comparison: Menthol-Preferring Smokers vs Non-Menthol Preferring Smokers; Least square means and standard errors were calculated to describe the patterns of means for each outcome. Effect slices were tested to explain significant interactions in the models. Pairwise comparisons of least square means were used to describe significant main effects; Test type: Other; p < .0001, Mixed Models Analysis; Mean Difference (Net) = .9436

ADVERSE EVENTS:
Time Frame: 4 hours
Description: The Systematic Assessment for Treatment Emergent Events (SAFTEE) was utilized to monitor adverse events.
  The Overall Number of Baseline Participants is not consistent with numbers provided any of the participant flow module due to analysis didn't include just number of completers but were analyzed by Day. (Adaptation, Day 1, Day 2 and Day 3)
Groups:
- Menthol-Preferring Smokers; Non-Menthol Preferring Smokers: Each subject in this arm received a random sequence of 3 different inhaled menthol conditions (3.2% menthol, 0.5% menthol and tobacco-flavor only (0.0% menthol)) across 3 test sessions (a single menthol condition for each test session). In each test session, a random order of one saline, and 2 nicotine (0.25 mg and 0.5 mg /70 kg) infusions were given one hour apart, concurrent with the randomized menthol inhalation condition.
Arm/Group | Menthol-Preferring Smokers | Non-Menthol Preferring Smokers
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/25
Other Adverse Events (participants affected / at risk) | 0/32 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT02102100/Prot_000.pdf